CLINICAL TRIAL: NCT05335317
Title: Study of the Efficiency and Safety of Low-Intensity Neodymium Laser Radiation With a Nanosecond Pulse Duration for Treatment of the Vaginal Walls Atrophic Changes
Brief Title: Treatment of Vaginal Atrophy With Low Intensity Nanosecond Neodymium Laser
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MeLSyTech, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TVALINNL-2019
Record Dates: First submitted 2022-04-13; First posted 2022-04-19 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Postmenopausal Period; Vaginal Atrophy; Vaginal Prolapse
Keywords: Vaginal Atrophy; Vaginal Prolapse; Neodymium Laser; Laser Treatment; Nanosecond; Laser; Vaginal; Postmenopausal
MeSH Terms: conditions — Uterine Prolapse | interventions — Laser Therapy; Vaginal Smears; Tomography, Optical Coherence; Biopsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The treatment method cannot be hidden from the participants and the researcher because of the very different method of treatment: laser treatment and the use of local hormones on their own. However, the specialists involved in the study (cytologist and ultrasound specialist) will not know which group the participant belongs to. The researcher will refer participants (or their materials) to these specialists, indicating their name and visit number. The Researcher will keep a document matching the participant's name and number.
  The conversation will be held with participants. The participant must not disclose his group when visiting an ultrasound specialist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Laser Treatment (Experimental): Laser treatment of the vagina, vulva, and paraurethral region with a "Magic Max" laser ("Magic Gyno"). In total, three procedures will be performed with an interval of 4-6 weeks.
  During the procedure, the following sequence of actions will be performed: 1st Stage - vaginal processing with a conical mirror handpiece, 2nd Stage - vaginal processing with a corner mirror handpiece, 3d Stage - external vulva and paraurethral region processing with a switched beam diameter handpiece.
  Interventions: Device: Laser Treatment; Diagnostic Test: Сlinical blood analysis; Diagnostic Test: Сlinical urine test; Diagnostic Test: Vaginal smear; Diagnostic Test: Cervical oncocytology test.; Diagnostic Test: Extended colposcopy; Diagnostic Test: Pelvic ultrasound; Other: King's Health Questionnaire; Diagnostic Test: Vaginal Health Index; Diagnostic Test: Ultrasound investigation; Diagnostic Test: Perineometry; Diagnostic Test: Optical coherence tomography; Diagnostic Test: Biopsy; Diagnostic Test: Femoflor screen
- Topical hormone (Active Comparator): Local hormone therapy with estriol. The course of treatment will be of 2 weeks of daily use, and then a maintenance therapy, when the suppository will be used of 2 times a week for 1.5-2 months to prevent symptoms.
  Interventions: Drug: Topical hormone estriol; Diagnostic Test: Сlinical blood analysis; Diagnostic Test: Сlinical urine test; Diagnostic Test: Vaginal smear; Diagnostic Test: Cervical oncocytology test.; Diagnostic Test: Extended colposcopy; Diagnostic Test: Pelvic ultrasound; Other: King's Health Questionnaire; Diagnostic Test: Vaginal Health Index; Diagnostic Test: Ultrasound investigation; Diagnostic Test: Perineometry; Diagnostic Test: Femoflor screen
- No treatment (Other): Participants without vaginal atrophy (no complaints of vaginal health and a vaginal health index greater than 20) and not receiving any treatment.
  Interventions: Diagnostic Test: Vaginal Health Index; Diagnostic Test: Optical coherence tomography; Diagnostic Test: Biopsy

INTERVENTIONS:
Device: Laser Treatment — Laser radiation is emitted by a series of pulses following each other through a pause. The duration of one pulse is 20-200 ns, the pause between pulses is 30 us. The energy of one pulse is about 1 mJ.
  General laser radiation parameters for 1st and 2nd stages are: beam with diameter of 4 millimeters (mm) scans treatment area by 4 circles with step of 2 mm (50% overlap), average power of 10-25 Watt (W), treatment time in one point of 1-10 seconds (s), treatment step of 5 mm (total handpiece length of 10 centimeter (cm), 20 treatment points along vagina), from 1 to 5 repetitions of total vagina treatment. General laser radiation parameters for 3d stage are: beam diameter of 6 mm, average power of 15-30 W, duration of ns-pulses packet of 100 milliseconds (ms), pause between packets of 50 ms, treatment duration up to 65 s, treatment in permanent motion with speed of 10-50 mm/s.
  The procedure is performed without anesthesia. The doctor always focuses on the participant's feeling of warmth.
  Arms: Laser Treatment
Drug: Topical hormone estriol — Estriol suppository ((17 beta)-estra-1,3,5 (10)-trien-3,17-diol). Active ingredient of 0.5 milligram in 1 suppository. Daily dose will be 1 suppository.
  Arms: Topical hormone
Diagnostic Test: Сlinical blood analysis — Taking blood from a vein for Clinical blood analysis (to include the participant in the study).
  Arms: Laser Treatment; Topical hormone
Diagnostic Test: Сlinical urine test — Urine sampling for Clinical urine test (to include the participant in the study).
  Arms: Laser Treatment; Topical hormone
Diagnostic Test: Vaginal smear — Vaginal smear for flora investigation (to include the participant in the study), immunocytochemical examination and cytology (to evaluate procedure efficiency).
  Arms: Laser Treatment; Topical hormone
Diagnostic Test: Cervical oncocytology test. — Cervical smear for oncocytology test (to include the participant in the study).
  Arms: Laser Treatment; Topical hormone
Diagnostic Test: Extended colposcopy — Extended colposcopy is performed under a microscope using a Lugol to determine external changes in the epithelium in order to determine atrophy and pathologies of the cervix and vaginal vault (dysplasia, erosion, cancer, etc.) (to include the participant in the study).
  Arms: Laser Treatment; Topical hormone
Diagnostic Test: Pelvic ultrasound — Pelvic ultrasound investigation to determine pathologies of the pelvic through a gynecological probe (to include the participant in the study).
  Arms: Laser Treatment; Topical hormone
Other: King's Health Questionnaire — The King's Health Questionnaire will be used to collect feedback on changes in the participants life quality (to evaluate procedure efficiency).
  Arms: Laser Treatment; Topical hormone
Diagnostic Test: Vaginal Health Index — Vaginal Health Index will be investigated by clinical examination for vaginal elasticity, vaginal secretions, epithelial mucous membrane, vaginal hydration. pH (potential of hydrogen) will be investigated by test-lines paper (to evaluate procedure efficiency).
Diagnostic Test: Ultrasound investigation — Ultrasound investigation with General Electric Voluson E8 Expert for assessing blood vessels (Doppler sonography) and vaginal wall thickness measurement (to evaluate procedure efficiency).
  Arms: Laser Treatment; Topical hormone
Diagnostic Test: Perineometry — Pressure force of vaginal walls measurement with IEASE device (to evaluate procedure efficiency).
  Arms: Laser Treatment; Topical hormone
Diagnostic Test: Optical coherence tomography — Optical non-invasive method of investigation vaginal mucus morphological and functional condition.
  Arms: Laser Treatment; No treatment
Diagnostic Test: Biopsy — Biopsy of the vaginal wall to assess the condition of the vaginal wall and compare the obtained data with the data of optical coherence tomography.
  Arms: Laser Treatment; No treatment
Diagnostic Test: Femoflor screen — Femoflor screen for the study of vaginal microbiocenosis, specifically for the detection of the pathogens, opportunistic flora and normal flora and their qualitative and quantitative evaluation (to include the participant in the study).
  Arms: Laser Treatment; Topical hormone

SUMMARY:
The aim of study is characteristic of changes in the vaginal wall after treatment of neodymium laser radiation with a wavelength of 1064 nm. To assess the condition of the vaginal walls before and after laser treatment, the following methods will be used: vaginal health index, perineometry, measurement of the vaginal wall thickness by ultrasound, Doppler sonography of the vaginal walls vessels, optical coherence tomography, biopsy, cytological and immunocytochemical methods. The King's Health Questionnaire will be used to collect feedback on changes in the participants life quality. Total up to 100 participants with and 20 participants without postmenopausal atrophy will be involved in the study. Participants will be divided into three groups: laser treatment (study group), topical hormones treatment (control group 1) and no treatment (control group 2) by 70, 30 and 20 participants in each group respectively. The time intervals between special tests and the tests themselves will be the same for all groups. Thus, a direct comparison between conventional treatment (topical hormones), laser treatment of the vaginal atrophy and normal condition without treatment will be made. The main hypothesis of the study is improvement in condition of the vaginal walls after laser treatment compared with the initial state of not less than thirty percent of participants, and improvement in condition on average compared with the control group.

DETAILED DESCRIPTION:
The principle of participant distribution into groups is the main method of treatment of postmenopausal vaginal atrophy. Total up to 100 participants with and 20 participants without postmenopausal atrophy will be involved in the study. Participants will be divided into three groups: laser treatment (study group), topical hormones treatment (control group 1), and no treatment (control group 2) by 70, 30, and 20 participants in each respectively.

The types of examination of each group are the same and include:

* General methods: clinical blood analysis, clinical urine test, vaginal smear for flora, femoflor screen (method is intended for the study of vaginal microbiocenosis), cervical oncocytology test, extended colposcopy, pelvic ultrasound.
* Special methods: filling out the questionnaire (King's Health Questionnaire), Vaginal Health Index, ultrasound for assessing blood vessels (Doppler sonography) and vaginal wall thickness, perineometry, optical coherence tomography (OCT), vaginal smear for immunocytochemical examination and cytology.

The TREATMENT PROCEDURE of this study is the laser treatment of the vagina and vulva with a "Magic Max" laser ("Magic Gyno" from August 2024) with subsequent monitoring.

Treatment Technique:

Laser treatment procedure will be carried out in three stages. In total, three procedures will be performed with an interval of 4-6 weeks. Three follow-up visits will follow: 1, 3 (mandatory) and 6 (optional) months after the last procedure.

During the procedure, the following sequence of actions will be performed:

1. st Stage - vaginal processing with a conical mirror handpiece,
2. nd Stage - vaginal processing with a corner mirror handpiece,
3. d Stage - external vulva and paraurethral region processing with a switched beam diameter handpiece.

Laser radiation is emitted by a series of pulses following each other through a pause. The duration of one pulse is 20-200 nanoseconds (ns), the pause between pulses is 30 microseconds (us). The energy of one pulse is about 1 millijoule (mJ). The procedure is performed without anesthesia. The doctor always focuses on the participant's feeling of warmth.

The CONTROL PROCEDURE. Local hormone therapy with estriol will be used as a therapeutic tool for the control group. The course of treatment will be of 2 weeks of daily use, and then a maintenance therapy, when the suppository will be used of 2 times a week for 1.5-2 months to prevent symptoms.

Participants of all groups will be tested with the general methods necessary to include the participant in the study at the first visit.

For the laser treatment group: Studies will be carried out using special methods and then laser treatment of the vagina and vulva and paraurethral region will be performed during the 2nd, 3d, and 4th visits. Studies with special methods only will be performed during the 5th (1 month after the last procedure), 6th (3 months after the last procedure), and 7th (6 months after the last procedure) visits.

For the control group 1 (hormonal treatment): Studies with special methods only will be performed during the 2nd, 3d, and 4th visits. Hormone therapy will begin from the 2nd visit. All subsequent visits will be carried out at the same time intervals as for the laser treatment group, using studies with special methods. The 3d visit will be in 4-6 weeks after the start of treatment, the 4th will be in 4-6 weeks after the 3d visit, the 5th - 1 month after the 4th, the 6th - 3 months after the 4th, the 7th - 6 months after the 4th.

Thus, a direct comparison between conventional treatment (topical hormones) and laser treatment of the vaginal atrophy will be made during the treatment, as well as on follow-up visits in 1, 3 and 6 months after the end of each type of treatment.

For the control group 2 Vaginal Health Index will be estimated only and OCT investigation with biopsy.

The study will be carried out with the participation of several clinics:

1. Privolzhsky Research Medical University (main scientific coordinator, information for participant recruiting),
2. State-Funded Healthcare Institution of the Nizhny Novgorod region "Nizhny Novgorod Regional Clinical Hospital named after N.A. Semashko" (location of laser equipment, laser treatment and participant consultation, special tests, collection of material for cytological and immunocytochemical analysis, recruiting),
3. Municipal Hospital №35 of the Soviet District of Nizhny Novgorod (cytological and immunocytochemical analysis),
4. State-Funded Healthcare Institution of the Nizhny Novgorod region "Municipal Clinical Hospital №29" (information for participant recruiting, general tests to include participants in the study),
5. LLC "Clinic of modern technologies "SADKO" (recruiting, general tests to include participants in the study, location of laser equipment, laser treatment and participant consultation, special tests, collection of material for cytological and immunocytochemical analysis),
6. Medical Center "Imidzh Lab" (information for participant recruiting, general tests to include participants in the study),
7. LLC "Tonus" (information for participant recruiting, general tests to include participants in the study).

All data obtained during the study will be transferred to the manufacturer of "MeLSyTech" Ltd.

Statistics

The analysis will be carried out both between groups of participants receiving different types of therapy (analysis of independent groups) and within groups at different time intervals (analysis of matched groups).

Before performing statistical analysis of the data, the distribution type of the variables will be assessed. To assess the normality of distribution for each variable, histograms of frequency distributions will be visually evaluated, indicators of skewness, kurtosis, and the D'Agostino-Pearson normality test will be used.

In addition to checking the type of distribution of variables, the equality of variances of the studied groups will be assessed using the methods of analysis of variance, in particular the Brown-Forsythe test.

Methods of descriptive analysis will be used depending on the type of distribution of the variable. With a normal distribution, the mean (M) and standard deviation (SD) will be calculated. In case of an nongaussian distribution, the median (Me) and interquartile range will be calculated. Different algorithms of statistical analysis will be applied depending on the type of distribution of variables.

Comparison of the paired and unpaired groups with a normal distribution, in case of the equality of the variances, will be carried out by the methods of analysis of variance ANOVA. Comparison of groups in pairs will be performed using the post-hoc method of posterior multiple comparisons (Tukey test).

Comparison of groups in which variables do not follow the normal distribution will be carried out using the methods of nonparametric analysis of variations: the Kruskal-Wallis test (ANOVA tests) for independent groups and the Friedman test for matched groups. Dunn's multiple comparison test will be used to assess intergroup differences.

Before assessing intergroup differences, the initial samples (1 visit) will be analyzed for identity using ANOVA or nonparametric Kruskal-Wallis tests (depending on the type of data). In case of significant differences in the samples, the search and removal of extremely deviating values (outliers) will be carried out.

Differences will be considered statistically significant if the significance P values are <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age of 40-75 years, inclusive;
* Vaginal atrophy or 1st grade vaginal prolapse with atrophy, or lack of vaginal atrophy in case of control group 2;
* All participants have informed consent to conduct a course of procedures according to protocol, carry out follow-up visits, and conduct studies.

Exclusion Criteria:

* Age of under 40 and over 75 years old;
* History of oncological diseases;
* Active tuberculosis;
* Inflammatory diseases of the vulva and vagina including genital herpes in the acute stage;
* Urinary tract infections;
* Damage to the vaginal mucosa;
* Pregnancy;
* Tendency to photoallergy including taking photosensitizing drugs (diuretics, antihistamines, antipsychotics);
* Porphyria;
* Cardiac deficiency of 2-3 degrees;
* Chronic renal disease;
* Participants with greater than 1st grade vaginal prolapse;
* Women after childbirth up to 8 weeks;
* Participants who, according to the doctor, are not able to complete the study;
* Protocol non-compliance of laser exposure sessions;
* Voluntary refusal to participate in the study;
* Violation of recommendations for the management of the period after laser treatment;
* Adverse events that occurred during laser processing and research, and associated with them.
* The appearance of contraindications listed in the Exclusion criteria.

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-04-18 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Mean Change from Baseline of Vaginal Health Index Score | 2nd visit (before any treatment); 3d visit (4-6 weeks after 2nd visit); 4th visit (4-6 weeks after 3d visit) - the end of any treatment; 1 month after 4th visit, 3 months after 4th visit, and 6 months after 4th visit
  Vaginal Health Index will be investigated by clinical examination for vagina:
  A. Vaginal elasticity (Characteristic=Points: Non=1, Poor=2, Fair=3, Good=4, Excellent=5), B. Vaginal secretions (None=1; Sсant, thin yellow=2; Superficial, thin white=3; Moderate, thin white=4; Normal (white)=5), C. Epithelial mucous membrane (Petechiae noted before contact=1, Bleeding with light contact=2, Bleeds with scraping, Not friable thin epithelium=4, Normal=5), D. Vaginal hydration (None, surface inflamed=1, None, surface nod inflamed=2, Minimal=3, Moderate=4, Normal=5), E. pH (potential of hydrogen) will be investigated by test-lines paper (≥6.1=1, 5.6-6.0=2, 5.1-5.5=3, 4.7-5.0=4, ≤4.6=5).
  Score=A+B+C+D+E
Mean Change from Baseline of Periodic Acid Schiff Reaction Percentage in Vaginal Smear | 2nd visit (before any treatment); 3d visit (4-6 weeks after 2nd visit); 1 month after 4th visit (after the end of any treatment), 3 months after 4th visit
  Part of a cytological test. Histological preparation prepared by liquid-based cytology and stained according to the instructions of the Periodic Acid Schiff kit. The investigator counts 100 cells in field of view with 400x magnification and records the proportion of cells with diffuse and granular staining. Parameter will be measured in percentages (%).
Mean Change from Baseline of Resistive Index by Doppler Sonography | 2nd visit (before any treatment);1 month after 4th visit (after the end of any treatment), 3 months after 4th visit, and 6 months after 4th visit
  Measurement is a part of ultrasonography. Resistive Index will be measured with US-device. The Resistive Index (RI) is calculated by the following equation: RI = (PSV - EDV) / PSV, where PSV is peak systolic velocity and EDV is end-diastolic velocity, in relative units.

OTHER OUTCOMES:
Mean Change from Baseline of "General Health Perceptions" Score on the King's Health Questionnaire | 2nd visit (before any treatment); 3d visit (4-6 weeks after 2nd visit); 4th visit (4-6 weeks after 3d visit) - the end of any treatment; 1 month after 4th visit, 3 months after 4th visit, and 6 months after 4th visit
  Participants answer question:
  Q1. How would participant describe her health at the present? Answers = Points: Very good=1, Good=2, Fair=3, Poor=4, Very poor=5. Score = ((Score to Q1 - 1)/4) x 100
Mean Change from Baseline of "Incontinence Impact" Score on the King's Health Questionnaire | 2nd visit (before any treatment); 3d visit (4-6 weeks after 2nd visit); 4th visit (4-6 weeks after 3d visit) - the end of any treatment; 1 month after 4th visit, 3 months after 4th visit, and 6 months after 4th visit
  Participants answer question:
  Q2. How much do participant think her bladder problem affects her life? Answers = Points: Not at all=1, A little=2, Moderately=3, A lot=4. Score =((Score to Q2 - 1)/3) x 100
Mean Change from Baseline of "Role Limitations" Score on the King's Health Questionnaire | 2nd visit (before any treatment); 3d visit (4-6 weeks after 2nd visit); 4th visit (4-6 weeks after 3d visit) - the end of any treatment; 1 month after 4th visit, 3 months after 4th visit, and 6 months after 4th visit
  Participants answer questions:
  A. Does participant's bladder problem affect her household tasks? (cleaning, shopping etc) B. Does participant's bladder problem affect her job, or her normal daily activities outside the home? Answers = Points: Not at all=1, Slightly=2, Moderately=3, A lot=4. Score =(((Scores to Q 3A + 3B) - 2)/6) x 100
Mean Change from Baseline of "Physical Limitations" Score on the King's Health Questionnaire | 2nd visit (before any treatment); 3d visit (4-6 weeks after 2nd visit); 4th visit (4-6 weeks after 3d visit) - the end of any treatment; 1 month after 4th visit, 3 months after 4th visit, and 6 months after 4th visit
  Participants answer questions:
  A Does participant's bladder problem affect her physical activities (e.g. going for a walk, running, sport, gym etc)? B. Does participant's bladder problem affect her ability to travel? C. Does participant's bladder problem limit her social life? D. Does participant's bladder problem limit her ability to see and visit friends? Answers = Points: Not at all=1, Slightly=2, Moderately=3, A lot=4. Score =(((Scores to Q 4A + 4B) - 2)/6) x 100
Mean Change from Baseline of "Social Limitations" Score on the King's Health Questionnaire | 2nd visit (before any treatment); 3d visit (4-6 weeks after 2nd visit); 4th visit (4-6 weeks after 3d visit) - the end of any treatment; 1 month after 4th visit, 3 months after 4th visit, and 6 months after 4th visit
  Participants answer questions:
  A Does participant's bladder problem affect her physical activities (e.g. going for a walk, running, sport, gym etc)? B. Does participant's bladder problem affect her ability to travel? C. Does participant's bladder problem limit her social life? D. Does participant's bladder problem limit her ability to see and visit friends? Answers = Points: Not at all=1, Slightly=2, Moderately=3, A lot=4. [If 5C >/= 1] Score =(((Score to Q 4C + 4D + 5C) - 3)/9) X 100 [If 5C = 0] Score =(((Score to Q 4C + 4D) - 2)/6) x 100
Mean Change from Baseline of "Personal Relationships" Score on the King's Health Questionnaire | 2nd visit (before any treatment); 3d visit (4-6 weeks after 2nd visit); 4th visit (4-6 weeks after 3d visit) - the end of any treatment; 1 month after 4th visit, 3 months after 4th visit, and 6 months after 4th visit
  Participants answer questions:
  A. Does participant's bladder problem affect her relationship with her partner? B. Does participant's bladder problem affect her sex life? C. Does participant's bladder problem affect her family life? Answers = Points: Not Applicable=0, Not at all=1, Slightly=2, Moderately=3, A lot=4.
  [If 5A+5B >=2]Score =(((Scores to Q 5A + 5B) - 2)/6) x 100 [If 5A+5B =1] Score =(((Scores to Q 5A + 5B) - 1)/3) x 100 [If 5A+5B =0] Treat as missing value
Mean Change from Baseline of "Emotions" Score on the King's Health Questionnaire | 2nd visit (before any treatment); 3d visit (4-6 weeks after 2nd visit); 4th visit (4-6 weeks after 3d visit) - the end of any treatment; 1 month after 4th visit, 3 months after 4th visit, and 6 months after 4th visit
  Participants answer questions:
  A. Does participant's bladder problem make she feel depressed? B. Does participant's bladder problem make she feel anxious or nervous? C. Does participant's bladder problem make she feel bad about herself? Answers = Points: Not at all=1, Slightly=2, Moderately=3, Very much=4. Score =(((Score to Q 6A + 6B + 6C) - 3)/9) X 100
Mean Change from Baseline of "Sleep / Energy" Score on the King's Health Questionnaire | 2nd visit (before any treatment); 3d visit (4-6 weeks after 2nd visit); 4th visit (4-6 weeks after 3d visit) - the end of any treatment; 1 month after 4th visit, 3 months after 4th visit, and 6 months after 4th visit
  Participants answer questions:
  A. Does participant's bladder problem affect her sleep? B. Does participant's bladder problem make she feel worn out and tired ? Answers = Points: Never=1, Sometimes=2, Often=3, All the time=4. Score =(((Scores to Q 7A + 7B) - 2)/6) x 100
Mean Change from Baseline of "Severity Measures" Score on the King's Health Questionnaire | 2nd visit (before any treatment); 3d visit (4-6 weeks after 2nd visit); 4th visit (4-6 weeks after 3d visit) - the end of any treatment; 1 month after 4th visit, 3 months after 4th visit, and 6 months after 4th visit
  Participants answer questions:
  Do participant do any of the following? A. Wear pads to keep dry? B. Be careful how much fluid she drink? C. Change her underclothes because it gets wet? D. Worry in case she smell? Answers = Points: Never=1, Sometimes=2, Often=3, All the time=4. Score =(((Scores to Q 8A + 8B + 8C + 8D) - 4)/12) x 100
Mean Change from Baseline of "Bladder Problems" Score on the King's Health Questionnaire | 2nd visit (before any treatment); 3d visit (4-6 weeks after 2nd visit); 4th visit (4-6 weeks after 3d visit) - the end of any treatment; 1 month after 4th visit, 3 months after 4th visit, and 6 months after 4th visit
  Participants answer questions:
  What participant's bladder problems are and how much they affect participant? From the list below participant chooses only those problems that she have at present. Participant leave out those that don't apply to she.
  FREQUENCY: going to the toilet very often NOCTURIA: getting up at night to pass urine URGENCY: a strong and difficult to control desire to pass urine URGE INCONTINENCE: urinary leakage associated with a strong desire to pass urine STRESS INCONTINENCE: urinary leakage with physical activity eg. coughing, running NOCTURNAL ENURESIS: wetting the bed at night INTERCOURSE INCONTINENCE: urinary leakage with sexual intercourse WATERWORKS INFECTIONS BLADDER PAIN Answers = Scores: Omitted=0, A little=1, Moderately=2, A lot=3.
Mean Change from Baseline of Pressure at Rest with IEASE Device | 2nd visit (before any treatment);1 month after 4th visit (after the end of any treatment), 3 months after 4th visit, and 6 months after 4th visit
  Measurement is a part of perineometry. Pressure at rest will be measured with IEASE device as inner function, in millimeter of mercury column (mmHg). Participants will be asked to hold the IEASE device bulb in normal condition of vagina without added pressure.
Mean Change from Baseline of Maximum Pressure at Contraction with IEASE Device | 2nd visit (before any treatment);1 month after 4th visit (after the end of any treatment), 3 months after 4th visit, and 6 months after 4th visit
  Measurement is a part of perineometry. Maximum pressure at contraction will be measured with IEASE device as inner function, in millimeter of mercury column (mmHg). Participants will be asked to hold the IEASE device bulb with maximum pressure they can.
Mean Change from Baseline of Constant Pressure Contraction Duration with IEASE Device | 2nd visit (before any treatment);1 month after 4th visit (after the end of any treatment), 3 months after 4th visit, and 6 months after 4th visit
  Measurement is a part of perineometry. Pressure at contraction will be measured with IEASE device as inner function, in millimeter of mercury column (mmHg).
  Participants will be asked to hold the IEASE device bulb for as long as they can with maximum pressure. The researcher will monitor the time from the beginning of contraction with maximum pressure to the moment when the pressure will decrease. Duration of constant pressure contraction will be measured with a stopwatch in seconds (s).
Mean Change from Baseline of Basal Cells Percentage in Vaginal Smear | 2nd visit (before any treatment); 3d visit (4-6 weeks after 2nd visit); 1 month after 4th visit (after the end of any treatment), 3 months after 4th visit
  Part of a cytological test. Vaginal smear is stained by Romanowsky. The investigator counts 100 cells in aliquot with 100x magnification and records the proportion of basal cells. Parameter will be measured in percentages (%).
Mean Change from Baseline of Parabasal Cells Percentage in Vaginal Smear | 2nd visit (before any treatment); 3d visit (4-6 weeks after 2nd visit); 1 month after 4th visit (after the end of any treatment), 3 months after 4th visit
  Part of a cytological test. Vaginal smear is stained by Romanowsky. The investigator counts 100 cells in aliquot with 100x magnification and records the proportion of parabasal cells. Parameter will be measured in percentages (%).
Mean Change from Baseline of Intermediate Cells Percentage in Vaginal Smear | 2nd visit (before any treatment); 3d visit (4-6 weeks after 2nd visit); 1 month after 4th visit (after the end of any treatment), 3 months after 4th visit
  Part of a cytological test. Vaginal smear is stained by Romanowsky. The investigator counts 100 cells in aliquot with 100x magnification and records the proportion of intermediate cells. Parameter will be measured in percentages (%).
Mean Change from Baseline of Superficial cells Percentage in Vaginal Smear | 2nd visit (before any treatment); 3d visit (4-6 weeks after 2nd visit); 1 month after 4th visit (after the end of any treatment), 3 months after 4th visit
  Part of a cytological test. Vaginal smear is stained by Romanowsky. The investigator counts 100 cells in aliquot with 100x magnification and records the proportion of superficial cells. Parameter will be measured in percentages (%).
Mean Change from Baseline of Keratinization Index in Vaginal Smear | 2nd visit (before any treatment); 3d visit (4-6 weeks after 2nd visit); 1 month after 4th visit (after the end of any treatment), 3 months after 4th visit
  Part of a cytological test. Vaginal smear is stained by Romanowsky. Parameter will be assessed in the five non-overlapping fields of view with magnification 400x as the ratio of the number of superficial cells to the number of all cells * 100. An average value will be calculated for each participant. Parameter will be measured in percentages (%).
Mean Change from Baseline of CK14 (Cytokeratin 14) Percentage in Vaginal Smear | 2nd visit (before any treatment); 3d visit (4-6 weeks after 2nd visit); 1 month after 4th visit (after the end of any treatment), 3 months after 4th visit
  Immunocytochemical examination. Histological preparation prepared by liquid-based cytology and stained according to the standard immunohistochemical protocol. Expression will be assessed in the 3-5 non-overlapping fields of view as the ratio of the number of positive-stained cells to the number of all cells * 100. An average value will be calculated for each participant. Parameter will be measured in percentages (%).
Mean Change from Baseline of Vaginal Wall Thickness by Ultrasound Scaled Image | 2nd visit (before any treatment);1 month after 4th visit (after the end of any treatment), 3 months after 4th visit, and 6 months after 4th visit
  Measurement is a part of ultrasonography. Thickness will be measured with US-device. The vaginal probe will be inserted into the posterior fornix of the vagina, the thickness of the vaginal wall will be determined by the distance between the inner surface of the mucosa and adventitia, in millimeters (mm).

CONTACTS AND LOCATIONS:
Overall Officials: Liya Z Sirotina, Principal Investigator — Privolzhsky Research Medical University
Locations (1):
- State-Funded Healthcare Institution of the Nizhny Novgorod region "Nizhny Novgorod Regional Clinical Hospital named after N.A. Semashko", Nizhny Novgorod, Russia

IPD SHARING:
Plan to Share IPD: Yes
The following data can be shared with researchers upon an official request:
  * The final version of the Study Protocol approved by the Local Ethics Committee;
  * Copies of anonymized filled Individual Registration Cards (IRC);
  * Informed Consent Form (ICF);
  * Clinical Study Report (CSR) and/or published article (if not contradict the rules and conditions of a journal);
  * Supplement files systematizing data.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: IPD can be shared with researchers starting 3 months after CSR or article publication for five years.
Access Criteria: IPD can be shared with researchers only upon an official request from researcher's affiliation institution in the letter form on organization's letterhead paper signed by an authorized person. Official request must be directed by e-mail to the contact person (Ksenia Shatilova, shatilova@melsytech.com). The letter must contain the request purpose and statement of internal IPD use as confidential information only.
  IPD will be shared after approval by CEO of "MeLSyTech" Ltd according to the company internal rules. A requester will be notified of the decision by official letter. Depending on the decision, a requester will receive a link to the repository, or a justified rejection.